CLINICAL TRIAL: NCT02075424
Title: Descriptive Study of Biological Stress and Perceived Stress in Call Regulation Operators and Doctors When Processing a Call at the Center 15
Brief Title: Descriptive Study of Biological Stress and Perceived Stress at the Center 15
Acronym: RegulStress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-02-CHRMT; 2013-A01725-40 (Other: ANSM)
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Physiological Stress; Psychological Stress
Keywords: stress; cortisol; emergency call center; hospital staff
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- salivery sampling by a biomnis swab (Experimental): Each call operator will have a series of salivary sampling taken when assigned to call reception, to the unit deployment station and to the assessment station.
  Only one sampling will occur to doctors who are assigned to a single workstation.
  Sampling will be taken every 15 minutes during one hour and half and one last sample will be taken 2 hours after the call For each participant, a serie of control-samples will be taken during a day off and during a security break.
  Interventions: Other: salivary sampling by a biomnis swab

INTERVENTIONS:
Other: salivary sampling by a biomnis swab — Each call operator will have a series of salivary sampling taken when assigned to call reception, to the unit deployment station and to the assessment station.
  Only one sampling will occur to doctors who are assigned to a single workstation.
  Sampling will be taken every 15 minutes during one hour and half and one last sample will be taken 2 hours after the call.
  To improve interpretation of the results, a series of control-samples will be taken among the call operators and doctors during a day off and not during a security break.
  There will be 4x8 samples taken for each call operator and 2x8 samples per doctor.
  They will also be frozen at a temperature of -4°C and sent to the laboratory of the CHR Metz Thionville.

SUMMARY:
The purpose of this study is to describe biological stress (cortisolemia) and perceived stress in Emergency Call Center Operators and Doctors while processing a center 15 call.

DETAILED DESCRIPTION:
Sample description : qualitative variables be expressed as percentages, numbers and 95% confidence intervals Quantitative variables will be expressed as means, standard deviations or medians, range, interquartile intervals Description of biological stress : it will be described by calculating the difference between the observed peek or peeks of cortisol ans the cortisol level measured at rest (means, standard deviations or medians, range, interquartile intervals) Description of perceived stress : the AVS will be described in terms of means and standard deviation Comparison of the peek-delta/base level of cortisol in the 3 different workstations of the call center operators according to the non parametrical Kruskall Wallis test. Same for the lengthof service of the call operator, the severity of the call and the status of the doctor The AVS score (perceived stress) will be compared to the peek-delta/base level of cortisol (biological stress) thanks to the Spearmann correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* medical and paramedical staff from the center 15 (call operators, emergency doctors and general practitioners)
* healthy volunteers having received the specific information letter regarding the sudy and having signed the clarified consent form
* healthy volunteers are affiliated to the french social welfare

Exclusion Criteria:

* chronic alcoholism
* women under oestroprogestative hormonal treatment
* high level athletes
* healthy volunteers under steroids treatment
* healthy volunteers suffering from a mental health related disorder
* fever on the day the sample is taken
* healthy volunteers with endocrine disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
biological stress by salivary cortisol secretion | every 15 minutes after the emergency call and during 2 hours

SECONDARY OUTCOMES:
perceived stress : VAS and SPPN questionnaire | VAS is assessed four times (once after each emergency call) during the first salivary sampling. SPPN once, on day 1, remote the emergency call (within the hourspreceding or following the emergency call)
  SPPN : Negative and Positive Professional Stress, before the first salivary sampling.
  VAS : Visual Analogic Scale,

CONTACTS AND LOCATIONS:
Overall Officials: Michel Aussedat, MD, Principal Investigator — Centre Hospitalier Régional Metz-Thionville
Locations (1):
- Centre Hospitalier Régional Metz Thionville, Metz, France

REFERENCES:
- [Background] Weibel L, Gabrion I, Aussedat M, Kreutz G. Work-related stress in an emergency medical dispatch center. Ann Emerg Med. 2003 Apr;41(4):500-6. doi: 10.1067/mem.2003.109. PMID 12658250
- [Background] Nakajima Y, Takahashi T, Shetty V, Yamaguchi M. Patterns of salivary cortisol levels can manifest work stress in emergency care providers. J Physiol Sci. 2012 May;62(3):191-7. doi: 10.1007/s12576-012-0197-8. Epub 2012 Feb 19. PMID 22350686
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychobiological research: an overview. Neuropsychobiology. 1989;22(3):150-69. doi: 10.1159/000118611. PMID 2485862
- [Background] Hellhammer DH, Wust S, Kudielka BM. Salivary cortisol as a biomarker in stress research. Psychoneuroendocrinology. 2009 Feb;34(2):163-171. doi: 10.1016/j.psyneuen.2008.10.026. Epub 2008 Dec 18. PMID 19095358
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychoneuroendocrine research: recent developments and applications. Psychoneuroendocrinology. 1994;19(4):313-33. doi: 10.1016/0306-4530(94)90013-2. PMID 8047637